CLINICAL TRIAL: NCT00956124
Title: Autofluorescence in Uveitic and Diabetic Macular Edema
Status: Withdrawn | Type: Observational
Why Stopped: Technical issue
Sponsor: St. Franziskus Hospital (Other)
Responsible Party: Principal Investigator, Carsten Heinz, Head of Department, St. Franziskus Hospital
Other Study IDs: 2009-017-f-S
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Uveitis; Macular Edema
MeSH Terms: conditions — Uveitis; Macular Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- uveitic patients
- patients with diabetes

SUMMARY:
The aim of this study is to determine whether fundus autofluorescence and macular pigment distribution in inflammatory and diabetic macular edema are altered.

DETAILED DESCRIPTION:
After macular pigment measuring we will perform fundus autofluorescence, fluorescein angiography and optical coherence tomography. any associations of macular pigment distribution and fundus autofluorescence with macular anatomic features are analyzed. primary outcome measure is the macular pigment distribution in patients with altered fundus autofluorescence. Furthermore we will compare the findings between diabetic and inflammatory edema.

ELIGIBILITY:
Inclusion Criteria:

* patients with diabetic or uveitis macular edema

Exclusion Criteria:

* children patients with known allergy to fluorescein

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with uveitis or diabetes
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology at St Franziskus Hospital, Münster, North-Rhine-Westfalia, Germany